CLINICAL TRIAL: NCT05288010
Title: CANPAIN Feasibility Study: Evaluating the Feasibility of Subsequently Undertaking a Pragmatic Real World Trial Investigating CBMP in Chronic Pain Patients
Brief Title: CANPAIN Feasibility Study Pragmatic Real World Trial Investigating CBMP in Chronic Pain Patients
Acronym: CANPAIN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Harley Street (CPC) Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 304548
Record Dates: First submitted 2022-02-22; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Chronic Pain
Keywords: Cannabis; Whole Flower Cannabis
MeSH Terms: conditions — Chronic Pain; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: Treatment with cannabis via an inhalation device in addition to standard of care chronic pain treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Group (Other): Patients of the clinic receiving cannabis treatment for non cancer chronic pain, who have been invited to join the study and have agreed and consented to join study.
  Interventions: Combination Product: Cannabis

INTERVENTIONS:
Combination Product: Cannabis — The provision of whole flower cannabis via an inhalation device in addition to standard of care chronic pain treatment.

SUMMARY:
The CANPAIN study has been devised to evaluate the efficacy and safety of a defined cannabis based medicinal product (CBMP) delivered by inhalation to patients with non cancer chronic pain attending a private clinic. CANPAIN is a pragmatic non-randomised, non-blinded real-world trial of the safety, tolerability and effectiveness of a cannabis based medicinal product (CBMP) for the treatment of chronic non-cancer pain compared against matched controls receiving standard of care pain management. CANPAIN will run for 3 years with a minimal planned sample size of 5000 participants per group who have completed at least 12 months of treatment. CANPAIN will be an MHRA and REC approved study. (See Appendix 1 of the Feasibility Study for the full draft protocol of the CANPAIN Study)

Prior to commencing the CANPAIN study, the sponsor proposes to conduct a feasibility study. This study will aid in establishing likely rates of patient recruitment, duration of participant enrolment in the study, the demographic and geographic spread of patients, patient acceptability of data collection and identify any issues with technological and drug delivery logistics.

DETAILED DESCRIPTION:
The feasibility study will be based within a private clinic setting and will only involve existing patients of the clinic. The treatment regime, tests that the patients are required to take, the clinical information they are required to provide, and the informed consent required for treatment, will all follow the clinical protocol. The sponsor wishes to assess the feasibility of conducting the study within the private clinic to aid a future submission to Oxford A REC of the CANPAIN study.

The feasibility study will be conducted over a 3-month period with a minimum target recruitment number of 100 patients. Feasibility will be assessed through 3 distinct domains: Recruitment and patient experience, medication logistics and data management.

Patient experiences (part of domain 3) will be captured using comment forms, requesting feedback on ease of onboarding, ease of answering questionnaires, evidence of questionnaire fatigue and their satisfaction of service.

ELIGIBILITY:
Inclusion Criteria:

1. A consented patient at the clinic;
2. Male or female 18-85 years old;
3. Diagnosed with chronic non-cancer pain;
4. Is currently receiving standard of care but still has pain, has completed standard of care pain treatment, does not want standard of care treatment, or standard of care is contraindicated. An inadequate response is defined as the subject receiving standard analgesic agents and still has pain, has unpleasant side effects or wishes to reduce their intake of standard of care analgesic agents, e.g. a subject receiving opioids who wishes to dose reduce in light of the "opioid crisis";
5. Despite being on or having received standard of care and has still pain (>3 on the Pain NRS); and
6. Signed and dated consent form from the patient.

Exclusion Criteria:

1. Pregnant or lactating females or females who are planning a pregnancy during the study;
2. Positive pregnancy test at time of joining the clinic;
3. Major organ failure, renal, lung or liver failure;
4. Participants having active liver disease or unexplained persistent elevation of serum transaminases > 3 times the upper limit of normal;
5. Participants with a creatinine clearance < 60mL/min;
6. History of cardiac or respiratory failure;
7. History of recent myocardial infarction or poorly controlled ischaemic heart disease;
8. Severe respiratory disease (e.g., GOLD 3 for COPD or asthmatics requiring high doses of oral corticosteroids);
9. History or presence of alcohol or substance abuse, including analgesics used as standard of care;
10. Participation in a clinical trial of an investigational medicinal product;
11. With any known or suspected history or family history of schizophrenia, or other psychotic illness; history of severe personality disorder or other significant psychiatric disorder disorders other than depression associated with their underlying condition;
12. Known hypersensitivity to cannabis or allergy to cannabis or CBMP; and
13. Currently taking cannabis and does not agree to a 3 week wash out period.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Experience | 3 months
  Assess rate of recruitment to the clinic. Measure time taken to recruit the first 100 patients from time of first patient in study until end of study. This will be measured using an electronic patient record which will record the date each patient entered and left the study.
Duration of Time in Study | 3 months
  Assess the number/proportion of patients that cease treatment at the Clinic. Measure the average time all patients remained in the study. This will be measured using an electronic patient record which will record the date each patient entered and left the study.
Questionnaire Compliance | 3 months
  Assess the number of patients that complete all questionnaires required. Measure the percentage of patients that completed all questionnaires required as part of the study.
Safety Questionnaire Results | 3 months
  Assess the number of patients that experience safety issues. Report the number of patients that recorded a score of 5 or more on the NRS tolerability questionnaire, in any of the safety questions.
Medication Logistics | 3 months
  Assess the timeliness and efficiency of CBMP delivery to the patient. Record average time taken for medication to reach patients after prescription has been completed using the shipping data from the pharmacy and the receipt date by the patient from the courier.
Device Experience | 3 months
  Assess the presence of issues with the usability of the inhalation device. Record number of patients that had issues with using the device from the comments questionnaire and from emails and phone calls to the study site.
Onboarding Experience | 3 months
  Ease of onboarding. Report from comments questionnaire and email and phone interactions with study site number of patients that had difficulties with registering with the clinic and entering into the study.
Questionnaire Logistics and Satisfaction | 3 months
  Ease of answering questionnaires. Record the number of patients that had problems with accessing or filling in the questionnaires from comments questionnaire and email and phone interactions with the study site.
Questionnaire Fatigue | 3 months
  Evidence of questionnaire fatigue. Report on the number of people that did not complete all questionnaires or did not complete them correctly or who complained about the number of questionnaires and questions in each questionnaire from the comments form and emails and phone calls to study site.
Patient Satisfaction with Service | 3 months
  Patients are required to fill out a Feedback Questionnaire which has a number of questions within it regards the service provided. Patients are required to rate the answers to these questions as Excellent, Good, Fair or Poor. The percentage of patients recording Excellent, Good, Fair and Poor will be calculated and tabulated and reported on.

SECONDARY OUTCOMES:
Demographic | 3 months
  Assess the socio-economic status and geographic origin of patients. Report on the number of patients by postcode to get an impression of socio-economic and demographic spread of the patients.
Conversion to Registration | 3 months
  Assess the number of enquiries to webpage and completion of registration forms. Report on the number of visits to the study site website and what percentage of these lead to a registration form being completed by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Shaw Sorooshian, MB ChB, Principal Investigator — LVL Health
Locations (1):
- LVL Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Summarised data will be made available via this site and peer review publications

DOCUMENTS (1):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT05288010/Prot_000.pdf